CLINICAL TRIAL: NCT04370704
Title: A Phase 1-2 Study of Combination Therapy With INCMGA00012 (Anti-PD-1), INCAGN02385 (Anti-LAG-3), and INCAGN02390 (Anti-TIM-3) in Participants With Select Advanced Malignancies
Brief Title: Study of Combination Therapy With INCMGA00012 (Anti-PD-1), INCAGN02385 (Anti-LAG-3), and INCAGN02390 (Anti-TIM-3) in Participants With Select Advanced Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCAGN 2385-201; 2021-005775-39 (EudraCT Number)
Expanded Access: NCT06910137 (Available)
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Melanoma
Keywords: PD-1 Inhibitors; INCAGN02385; INCAGN02390; INCMGA00012; Retifanlimab
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1 Part 1 (Experimental): Part 1 will confirm the safety of INCAGN02385 and INCAGN02390 when used in combination. INCAGN02385 will be administered first intravenously followed by INCAGN02390.
  Interventions: Drug: INCAGN02385; Drug: INCAGN02390
- Phase 1 Part 2 (Experimental): Part 2 will confirm the safety of the triple combination of INCAGN02385 + INCAGN02390 + INCMGA00012, following confirmation of the safety of the doublet in Part 1. INCAGN02385 will be administered first intravenously followed by INCAGN02390 and INCMGA00012.
  Interventions: Drug: INCAGN02385; Drug: INCAGN02390; Drug: INCMGA00012.
- Phase 2 Cohort A (Experimental): Phase 2 will determine preliminary efficacy and proof of concept for the combination of INCAGN02385 + INCAGN02390 + INCMGA00012. INCAGN02385 will be administered first intravenously followed by INCAGN02390 and INCMGA00012
  Interventions: Drug: INCAGN02385; Drug: INCAGN02390; Drug: INCMGA00012.
- Phase 2 Cohort B (Experimental): Phase 2 will determine preliminary efficacy and proof of concept for the combination of INCAGN02385 + INCAGN02390 + INCMGA00012. INCAGN02385 will be administered first intravenously followed by INCAGN02390 and INCMGA00012
  Interventions: Drug: INCAGN02385; Drug: INCAGN02390; Drug: INCMGA00012.
- Phase 1 Part 3 (Experimental): Part 1 will confirm the safety of INCAGN02385 + INCAGN02390 + INCMGA00012 when used in combination.
  Interventions: Drug: INCAGN02385; Drug: INCAGN02390; Drug: INCMGA00012.
- Phase 1 Part 4 (Experimental): Part 1 will confirm the safety of INCAGN02385 + INCAGN02390 + INCMGA00012 in combination.
  Interventions: Drug: INCAGN02385; Drug: INCAGN02390; Drug: INCMGA00012.

INTERVENTIONS:
Drug: INCAGN02385 — INCAGN02385 administered intravenously
Drug: INCAGN02390 — INCAGN02390 administered intravenously
Drug: INCMGA00012. — INCMGA00012 administered intravenously
  Arms: Phase 1 Part 2; Phase 1 Part 3; Phase 1 Part 4; Phase 2 Cohort A; Phase 2 Cohort B

SUMMARY:
The study will determine Recommended Phase 2 Dose for all study drugs, based on the safety and tolerability of the following combinations: INCAGN02385 + INCAGN02390 and INCAGN02385 + INCAGN02390 + INCMGA00012.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 Parts 1-4): Participants with locally advanced or metastatic solid tumors (locally advanced disease must not be amenable to resection with curative intent) that have failed available therapies, including anti-PD-(L)1 therapy if applicable, that are known to confer clinical benefit, or who are intolerant to, or ineligible for standard treatment. Prior anti-PD-(L)1 therapy should not have been discontinued because of intolerance.
* Phase 2, Cohort A:

  1. Participant with histologically confirmed unresectable/metastatic melanoma, whose disease failed prior anti-PD-(L)1 therapy (alone or as part of a combination) and meeting one of the following criteria:

     * Participant who failed prior adjuvant anti-PD-(L)1 therapy for resectable melanoma must have received prior anti-PD-(L)1 for ≥ 6 weeks and experienced disease progression while still on active adjuvant therapy containing anti-PD-(L)1, or participant who had early relapse occurring < 24 weeks after end of adjuvant anti-PD-(L)1 therapy. Progressive disease must be ascertained by confirmatory biopsy collected at baseline.
     * Participant whose unresectable/metastatic disease progressed while on or within < 24 weeks of completion of anti-PD-(L)1 for inresectable/metastatic melanoma. Progressive disease must have been confirmed by imaging ≥ 4 weeks after evidence of initial disease progression.
  2. Participant must have received no more than 2 prior lines of therapy for melanoma and at least one prior regimen must have contained anti-PD-(L)1 therapy (alone or as part of a combination) either in the adjuvant and/or advanced/metastatic setting.
  3. Participants must have had known BRAF V600 mutation status per local institutional testing standards.
  4. Participants must have fresh biopsy available after completing prior PD-(L)1 therapy or be willing and able to safely undergo pretreatment tumor biopsies (core or excisional). Determination of whether participants can safely undergo biopsy should be made by the treating physician in consultation with the individual performing the biopsy.
  5. Participant must have at least 1 measurable tumor lesion per RECIST v1.1.
* Phase 2, Cohort B:

  1. Participant with previously untreated, histologically confirmed Stage III (unresectable) or IV melanoma per the American Joint Committee on Cancer v8 staging system.
  2. Participants must not have had prior systemic anticancer therapy for unresectable or metastatic melanoma.
  3. Participants must have had known BRAF V600 mutation status per local institutional testing standards.
  4. Participants must have fresh biopsy available or be willing and able to safely undergo pretreatment tumor biopsies (core or excisional). Determination of whether participants can safely undergo biopsy should be made by the treating physician in consultation with the individual performing the biopsy.
* Phase 2 (Cohorts A and B): Participant must have at least 1 measurable tumor lesion per RECIST v1.1.
* ECOG performance status 0 or 1.
* Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

* Laboratory and medical history parameters outside the protocol-defined range.
* Known hypersensitivity or severe reaction to any component of the study drugs or formulation components ) within 14 days before study Day 1.
* Participant who had prior treatment with a LAG-3 or TIM-3 targeted agent.

Phase 1: (Parts 1-4):

* Receipt of anticancer medications or investigational drugs within the following intervals before the first administration of study treatment:

  1. ≤28 days or 5 half-lives (whichever is longer) before the first dose for all other investigational agents or devices. For investigational agents with long half-lives (eg, > 5 days), enrollment before the fifth half-life requires medical monitor approval.
  2. Administration of colony-stimulating factors (including granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 14 days before study Day 1.
* Phase 2:
* Cohort A: Participant who has discontinued anti-PD-(L)1 therapy due to toxicity or other reasons unrelated to toxicity, then subsequently experienced disease progression.
* Cohort A: Participant who had experienced objective response (PR/CR) and had stopped anti-PD-(L)1 therapy due to maximal benefit.
* Cohort A: Participant with multiple metastases that achieved mixed tumor response to prior anti-PD-(L)1 therapy (such as isolated progressive lesion in a context of PR/CR or SD for other lesions) or achieved overall disease progression based only on a single new lesion.
* Cohort B: Participant who has or has had uveal melanoma.
* Receipt of anticancer therapy (immunotherapy, chemotherapy, targeted therapy or hormonal therapy) within 21 days of the first administration of study treatment, with the exception of localized radiotherapy.
* Palliative radiation therapy administered within 1 week of first dose of study treatment or radiation therapy in the thoracic region that is > 30 Gy within 6 months of the first dose of study treatment.
* If participant received major surgery, then they must have recovered adequately from toxicities and/or complications from the intervention before starting study treatment.
* Treatment-related toxicity related to prior therapy that has not recovered to ≤ Grade 1 (with the exception of alopecia and anemia not requiring transfusional support), unless approved by the medical monitor.
* History of immune-related toxicity during prior checkpoint inhibitor therapy for which permanent discontinuation of therapy is recommended (per product label or consensus guidelines), OR any immune-related toxicity requiring intensive or prolonged immunosuppression to manage (with the exception of endocrinopathy that is well controlled on stable dose of replacement hormones such as hypothyroidism or adrenal insufficiency, or Grade 3 rashes that resolved with topical therapy or asymptomatic lipase elevations that do not require treatment interruption or uveitis that resolved with steroid drops).
* Has an active autoimmune disease requiring systemic immunosuppression with corticosteroids (> 10 mg/day of prednisone or equivalent) or immunosuppressive drugs within 14 days before the first dose of study treatment.
* Receiving chronic systemic corticosteroids (> 10 mg/day of prednisone or equivalent).
* Active infections requiring systemic antibiotics, or antifungal or antiviral treatment within 7 days before first dose of study treatment.
* History of organ transplant, including allogeneic stem cell transplantation.
* Evidence of interstitial lung disease or active, noninfectious pneumonitis.
* Known active HBV or HCV infection or risk of reactivation of HBV or HCV.
* Participants who are known to be HIV-positive .
* Known active brain or CNS metastases including carcinomatous meningitis.
* Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy after treatment with curative intent.
* Participants with impaired cardiac function or clinically significant cardiac disease
* History or presence of an abnormal ECG that, in the investigator's opinion, is clinically meaningful.
* Women who are pregnant or breastfeeding.
* Receipt of a live vaccine within 30 days of planned start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Phases 1 & 2: Participants with treatment-emergent adverse events (TEAEs) | 28 days after end of study approximately 24 months
  TEAE is defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug
Phase 2 Cohort A and B: Objective Response Rate (ORR) | Every 8 weeks for first 12 months, and every 12 weeks until disease progression; approximately 24 months
  Defined as the percentage of participants having a Complete Response or Partial Response, will be determined by investigator assessment of radiographic disease assessments per RECIST v1.1.
Phase 2 Cohort A and B: Duration of Response (DOR) | Every 8 weeks for first 12 months, and every 12 weeks until disease progression; approximately 24 months
  Defined as the time from earliest date of disease response (CR or PR) until earliest date of disease progression, as determined by investigator assessment of radiographic disease per RECIST v1.1, or death from any cause, if occurring sooner than progression.
Phase 2 Cohort A and B: Disease Control Rate (DCR) | Every 8 weeks for first 12 months, and every 12 weeks until disease progression; approximately 24 months
  Defined as percentage of participants having CR, PR, or SD as best on-study response.
Phase 2 Cohort A and B: Progression-free Survival (PFS) | Every 8 weeks for first 12 months, and every 12 weeks until disease progression; approximately 24 months
  Defined as the time from date of first dose of study treatment until the earliest date of disease progression, as determined by investigator assessment of objective radiographic disease per RECIST v1.1

SECONDARY OUTCOMES:
Phase 1 : Objective Response Rate | Every 8 weeks for first 12 months, and every 12 weeks until disease progression; aprroximately 24 months
  Defined as the percentage of participants having a Complete Response or Partial Response, will be determined by investigator assessment of radiographic disease assessments per RECIST v1.1.
Phase 1 : Progression Free Survival | Every 8 weeks for first 12 months, and every 12 weeks until disease progression; aprroximately 24 months
  Defined as the time from date of first dose of study treatment until the earliest date of disease progression, as determined by investigator assessment of objective radiographic disease per RECIST v1.1.
Phase 1: Disease Control Rate (DCR) | Every 8 weeks for first 12 months, and every 12 weeks until disease progression; approximately 24 months
  Defined as percentage of participants having CR, PR, or SD as best on-study response

CONTACTS AND LOCATIONS:
Locations (17):
- United States (12):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - H Lee Moffitt Cancer Center and Research, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Cancer Center For Blood Disorders A Division of American Oncology Partners P.A, Bethesda, Maryland
  - Washington University, St Louis, Missouri
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Nyu Langone Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Carolina Bio Oncology, Huntersville, North Carolina
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Washington-Seattle Cancer Care Alliance, Seattle, Washington
- Australia (5):
  - Melanoma Institute Australia, Wollstonecraft, New South Wales
  - Greenslopes Private Hospital, Brisbane, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - One Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency